CLINICAL TRIAL: NCT02929381
Title: A Prospective Randomized Clinical Trial to Assess the Utility of Advanced Endoscopic Imaging and the Impact of New Technologies on Quality in Colonic Examinations
Brief Title: Advanced Endoscopic Imaging in Colonoscopy
Acronym: AEI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miroslaw Szura (Other)
Collaborators: Specialist Diagnostic and Therapeutic Center MEDICINA (Unknown); Jagiellonian University (Other)
Responsible Party: Sponsor-Investigator, Miroslaw Szura, Associate Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ADVANCED ENDOSCOPIC IMAGING
Record Dates: First submitted 2016-09-30; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Polyps; Neoplasms
Keywords: Narrow Band Imaging; Colorectal Cancer Screening; Colonoscopy; Responsive Insertion Technology; Near Focus
MeSH Terms: conditions — Polyps; Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Innovative colonoscopy (Experimental): Innovative colonoscopy performed using narrow band imaging and dual focus function (NBI + Dual Focus)
  Interventions: Device: Innovative colonoscopy (Olympus CF-HQ190L, NBI + Dual Focus)
- Conventional colonoscopy (Active Comparator): Conventional colonoscopy performed without innovative techniques assessed in this study.
  Interventions: Device: Conventional colonoscopy (Olympus CF-H180DL)

INTERVENTIONS:
Device: Innovative colonoscopy (Olympus CF-HQ190L, NBI + Dual Focus) — NBI and Dual Focus options will be used to classify lesions according to Kudo and NICE classifications.
  Arms: Innovative colonoscopy
Device: Conventional colonoscopy (Olympus CF-H180DL) — Conventional colonoscopy performed without innovative techniques used in experimental arm.
  Arms: Conventional colonoscopy

SUMMARY:
The aim of the study is to evaluate the usefulness of high-tech endoscopy in clinical practice.

The important elements of this evaluation are:

* Evaluation of the character of neoplastic lesions in the colon based on different imaging techniques
* Verification of the endoscopic image with histopathologic descriptions
* Establishing the type of the lesion on the basis of Kudo and NICE classifications
* Comparison of the result of histopathological examination with the macroscopic type of the lesion
* Determination of the most advanced lesions (MAL)
* Comparison of the cecal intubation time
* Evaluation of the type of anesthesia used during colonoscopy
* Subjective assessment of the severity of pain according to VAS (visual analogue scale)
* Comparison of the accuracy of the location of lesions on the basis of endoscopic navigation
* Comparison of the total examination time
* Comparison of adenoma detection rate

DETAILED DESCRIPTION:
A total of 400 consecutive patients undergoing unsedated colonoscopy as a part of a national colorectal cancer screening program will be randomly assigned to innovative or conventional examination. Randomization will be based on computer-generated randomization lists. All patients will be blinded so they will not know which techniques will be used to assess lesions found in colon. In innovative colonoscopy group narrow band imaging (NBI) and Dual Focus (DF) function will be used to identify and classify all lesions according. to Kudo and NICE classification. Endoscopic biopsy samples will be taken from all lesions and in vivo endoscopic diagnosis will be compared with final histopathological result. Thus, sensitivity, specificity, diagnostic accuracy, predictive values, likelihood ratio and Youden index will be calculated. As secondary endpoints total examination time, cecal intubation rate and pain intensity (VAS) will be determined. This study will help to establish whether advanced imaging technologies used during colonoscopy may improve diagnostic possibilities and whether they prolong examination time or lead to increase of pain intensity afterwards.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* no previous abdominal surgery
* no colonoscopy during last 10 years

Exclusion Criteria:

* age < 40 and > 65 years
* large bowel resection in history
* colonoscopy performed during last 10 years
* contraindications for general anaesthesia
* ASA > IV
* pregnancy
* confirmed neoplastic disease
* cirrhosis (Child B or C) or ascites
* immunosuppressive therapy or steroids intake
* malabsorption syndrome
* IBD
* GI neoplastic disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of innovative colonoscopy | 1 year
  Diagnostic accuracy of innovative techniques used during colonoscopy (narrow band imaging and double focus option) will be assessed using StatSoft Statistica 10.0 software. All lesions will be classified acc. to NICE and Kudo classification during colonoscopy and results will be compared with histologic examination.

SECONDARY OUTCOMES:
Total examination time | 8-20 minutes
  Time of the whole procedure (from insertion of the colonoscope to removing of the whole instrument) will be compared in conventional and innovative colonoscopy.
Cecal intubation time | 5-15 minutes
  Time from insertion of colonoscope to visualisation of the coecum - always confirmed by a snapshot.
Pain intensity (VAS scale) | immediately after colonoscopy, 15 min, 30 min, 1 hour and 2 hours after the procedure
  Pain intensity will be assessed during and after each colonoscopy using the Visual Analogue Scale. It will be assessed immediately after colonoscopy, 15 min, 30 min, 1 hour and 2 hours after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslaw Szura, MD, PhD, Principal Investigator — Department of Experimental and Clinical Surgery, Jagiellonian University Medical College,; Artur Pasternak, MD, PhD, Study Chair — Department of Anatomy, Jagiellonian University Medical College
Locations (1):
- Specialist Diagnostic and Therapeutic Center MEDICINA, Krakow, Malopolska, Poland

REFERENCES:
- [Derived] Bogacki P, Gach T, Krzak J, Szura M. Panoramic colonoscopy in colorectal cancer screening - a randomized controlled trial. Wideochir Inne Tech Maloinwazyjne. 2021 Jun;16(2):289-296. doi: 10.5114/wiitm.2021.103922. Epub 2021 Feb 25. PMID 34136023